CLINICAL TRIAL: NCT00424346
Title: A 12-week, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group, Dose-finding Study to Evaluate the Efficacy, Safety and Tolerability of ACZ885 (Anti-interleukin-1beta Monoclonal Antibody) With Three Different Dose Regimens in Patients With Active Rheumatoid Arthritis Despite Stable Treatment With Methotrexate Including 76-week and 96-week Extensions
Brief Title: Efficacy, Safety and Tolerability of ACZ885 in Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CACZ885A2201; CACZ885A2201E1; CACZ885A2201E2; NCT00471198 (obsolete NCT alias); NCT00784628 (obsolete NCT alias)
Record Dates: First submitted 2007-01-17; First posted 2007-01-19 (Estimated); Results first posted 2013-06-19 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2013-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Active Rheumatoid Arthritis; anti-interleukin-1beta monoclonal antibody; methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Canakinumab 600 mg IV + 300 mg q2wk (Experimental): Participants received canakinumab 600 mg intravenous (IV) loading dose on Day 1 and 300 mg subcutaneous injections every 2 weeks (q2wk) for 12 weeks in the Core Phase. In the Extension Phase, participants received 300 mg canakinumab every 4 weeks subcutaneously, until a protocol amendment in January 2009 decreased the dose to 150 mg every 4 weeks.
  Interventions: Drug: Canakinumab
- Canakinumab 300 mg q2wk (Experimental): Participants received canakinumab 300 mg subcutaneous injections every 2 weeks (q2wk) for 12 weeks in the Core Phase. In the Extension Phase, participants received 300 mg canakinumab every 4 weeks subcutaneously, until a protocol amendment in January 2009 decreased the dose to 150 mg subcutaneous injection every 4 weeks.
  Interventions: Drug: Canakinumab
- Canakinumab 150 mg q4wk (Experimental): Participants received canakinumab 150 mg subcutaneous injections every 4 weeks (q4wk) for 12 weeks in the Core Phase. In the Extension Phase, participants received 300 mg canakinumab every 4 weeks subcutaneously, until a protocol amendment in January 2009 decreased the dose to 150 mg subcutaneous injection every 4 weeks.
  Interventions: Drug: Canakinumab
- Placebo (Placebo Comparator): Participants received placebo subcutaneous injections every 2 weeks for 12 weeks in the Core Phase. In the Extension Phase, participants received 300 mg canakinumab every 4 weeks subcutaneously, until a protocol amendment in January 2009 decreased the dose to 150 mg subcutaneous injection every 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Canakinumab
  Other Names: ACZ885
  Arms: Canakinumab 150 mg q4wk; Canakinumab 300 mg q2wk; Canakinumab 600 mg IV + 300 mg q2wk
Drug: Placebo
  Arms: Placebo

SUMMARY:
The 12-week core study was designed to evaluate risk-benefit of three subcutaneous dose regimens of ACZ885, added on to stable methotrexate (MTX) therapy (greater than or equal to 7.5 mg/week), compared to placebo in patients with active rheumatoid arthritis (RA). The study investigated the magnitude of effect as well as onset of effect for the different dose regimens.

The primary objective of the extension studies was to assess long-term safety and tolerability of canakinumab (ACZ885) in patients with active RA. CACZ885A2201E1 evaluated this objective in patients who had participated in the core study (CACZ885A2201) and CACZ885A2201E2 did the same in patients who completed the first extension study.

ELIGIBILITY:
Other protocol-defined inclusion/exclusion criteria may apply

CORE STUDY

Inclusion Criteria

Core Study Inclusion Criteria At Screening

1. Cooperative male or non-pregnant, non-lactating female patients at least 18 years of age who signed an informed consent before the initiation of any study procedure.
2. Diagnosis of rheumatoid arthritis (RA) classified by American College of Rheumatology (ACR) 1987 revised criteria and with symptoms for at least 3 months before randomization.
3. Functional status class I, II or III classified according to the ACR 1991 revised criteria.
4. Patients treated with methotrexate (MTX) at the maximum tolerated (≤25 mg/week) and stable dose of ≥7.5 mg/week for at least 12 weeks before randomization.
5. Patients who had failed any disease-modifying antirheumatic drugs (DMARDs) (including biologic agents and any DMARD used in combination with MTX) were allowed.
6. For patients with previous treatment of biological therapy, the following wash-out periods were required before randomization:

   * 3 days for Kineret™ (anakinra) - with a terminal half-life of 4 to 6 hours (s.c. route).
   * 4 weeks for Enbrel® (etanercept) - with a terminal half-life of 102 ± 30 hours (s.c.

   route).
   * 8 weeks for Remicade® (infliximab) - with a terminal half-life of 8.0-9. 5 days (intravenous (i.v.) infusion).
   * 12 weeks for Humira® (adalimumab) - with a terminal half-life of 10-20 days (average 2 weeks) (subcutaneous (s.c.) route).
   * 12 weeks for Orencia® (abatacept) - with a terminal half-life of 13.1 (8-25) days (i.v. infusion).
   * 26 weeks for any other biologic - or 10 half-lives, whichever was longer.
7. Patients who took systemic corticosteroids had to be on a stable dose of ≤10 mg/d prednisone or equivalent for at least 4 weeks before randomization.
8. Patients who were regularly taking non-steroidal anti-inflammatory drugs (NSAIDs) or COX-2 inhibitors or paracetamol/ acetaminophen as part of their RA therapy must have been on a stable dose for at least 4 weeks before randomization. Patients taking NSAIDs or COX-2 inhibitors or paracetamol/acetaminophen as needed within 2 weeks before randomization had to stop their medication at least 24 hours before an ACR visit (i.e. Visits 3, 7, 8, 10 and 12 [End of Study]). Patients taking folic acid supplementation had to be on stable dose for at least 4 weeks before randomization.
9. Patients with a history of immunization for Influenza (within past 12 months) and Pneumococcal vaccination (within 4 years) were included. If not already immunized, vaccination was completed when medically indicated (only during flu season for influenza) and such patients were included after approximately a 3 week window post-immunization to allow immunity to develop for vaccine.
10. Weight ≥45 kg and body mass index (BMI) <34.0
11. Women of non-child-bearing potential, defined as all women physiologically not capable of becoming pregnant.

Core Study Inclusion criteria At Baseline (Visit 3)

1. Disease activity criteria of ≥6 out of 28 tender joints and ≥6 out of 28 swollen joints.
2. One of the following also had to be present:

   1. High-sensitive C-Reactive Protein (hsCRP) concentration ≥10 mg/L
   2. Erythrocyte Sedimentation Rate (ESR) ≥28 mm/1st hr
   3. a. + b. based on screening values.

EXCLUSION

1. History of hypersensitivity to study drug or to molecules with similar structures.
2. Any therapy by intra-articular injections (e.g. corticosteroid) required for treatment of acute RA flare within 4 weeks before randomization.
3. Current use of DMARDs other than MTX. DMARDs included but were not limited to: biologic agents, thiolates (D-penicillamine, thiopronine), sulfasalazine, gold compounds, antimalarials, cyclosporine A, azathioprine, leflunomide, and alkylating agents such as cyclophosphamide.
4. If a patient had been discontinued from DMARDs, the patient should have been off the agent for at least 4 weeks, except leflunomide which was 8 weeks.
5. Patients with evidence of active pulmonary disease (e.g. tuberculosis, fungal diseases).
6. Donation or loss of 400 mL or more of blood within 8 weeks prior to dosing.
7. Who had a live vaccination within 12 weeks before randomization, or were planning to have one during the study and were not willing/able to postpone until study completion.
8. a) With bacterial, fungal or viral infections at the time of enrollment, including patients with evidence of human immunodeficiency virus (HIV) infection, hepatitis B and hepatitis C infection.

   b) History of a positive purified protein derivative (PPD) of tuberculin skin test without a follow-up of a negative chest X-ray.

   c) Patients requiring administration of antibiotics against latent tuberculosis, e.g. isoniazide.
9. Underlying metabolic, hematologic, renal, hepatic, infectious or gastrointestinal conditions which in the opinion of the investigator immunocompromised the patient and/or placed the patient at unacceptable risk for participation in an immunomodulatory therapy. In particular, clinical evidence or history of multiple sclerosis or other demyelinating diseases, or Felty's syndrome.
10. With significant medical problems, including but not limited to the following: uncontrolled hypertension (≥160/95 mmHg), congestive heart failure, type-I-diabetes(well controlled type-II-diabetes was allowed even when requiring insulin), thyroid disease (unless the patient was taking a stable dose of thyroid hormone for at least 12 weeks before randomization).
11. Other rheumatic diseases that could confound the evaluation of efficacy, including but not limited to primary fibromyalgia, ankylosing spondylitis, Lyme disease, adult juvenile RA, systemic lupus erythematosus, gout and pseudo gout, vasculitis, psoriatic arthritis, reactive arthritis, primary Sjoegren's Syndrome, and Behcet's Syndrome.
12. Any medical or psychiatric condition which, in the Investigator's opinion, would preclude the participant from adhering to the protocol or completing the study per protocol.
13. History of malignancy of any organ system, treated or untreated, within the past 5 years (with the exception of adequately treated basal cell carcinoma or squamous-cell carcinoma of the skin, carcinoma in situ of the cervix, colon polyps with non-invasive malignancy that have been removed).
14. Use of any investigational drug other than RA therapy and/or devices at the time of randomization, or within 30 days or 5 half- lives of randomization, whichever was longer.

STUDY EXTENSIONS

Extension Studies Inclusion Criteria:

1. Patients who completed the core CACZ885A2201 study may enter the first extension study upon signing informed consent. A patient is defined as completing the study if he/she completed the core CACZ885A2201 study up to and including Visit 12.
2. Patients who completed the first extension study, may enter the second.

Extension Studies Exclusion Criteria

1. Patients for whom continued treatment in the extension is not considered appropriate by the treating physician.
2. Patients who were non-compliant or who demonstrated a major protocol violation in the core CACZ885A2201 study.
3. Patients who discontinued from the core CACZ885A2201 study before Visit 12.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2006-11; Primary Completion 2008-09 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (12):
  - Pinnacle Research Group, Anniston, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Sun Valley Arthritis Center, Ltd, Peoria, Arizona
  - Catalina Pointe Arthritis & Rheumatology Specialists, Tucson, Arizona
  - Arthritis Center, Palm Harbor, Florida
  - Arthritis Research of Florida, Inc., Palm Harbor, Florida
  - The Arthritis Center, Springfield, Illinois
  - St. Louis Cener for Clinical Research, St Louis, Missouri
  - The Center for Rheumatology, Albany, New York
  - AAIR Research Center, Rochester, New York
  - Oregon Health Sciences University, Portland, Oregon
  - Tacoma Center for Arthritis Research, Tacoma, Washington
- Novartis, Vienna, Austria
- Novartis, Vilvoorde, Belgium
- Novartis, Dorval, Quebec, Canada
- Novartis, Nuremberg, Germany
- Novartis, Barcelona, Spain

REFERENCES:
- [Derived] Alten R, Gomez-Reino J, Durez P, Beaulieu A, Sebba A, Krammer G, Preiss R, Arulmani U, Widmer A, Gitton X, Kellner H. Efficacy and safety of the human anti-IL-1beta monoclonal antibody canakinumab in rheumatoid arthritis: results of a 12-week, Phase II, dose-finding study. BMC Musculoskelet Disord. 2011 Jul 7;12:153. doi: 10.1186/1471-2474-12-153. PMID 21736751

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 277 patients were randomized in core (CACZ885A2201): 71 were assigned to ACZ885 600 mg intravenous(iv) + 300 mg subcutaneous each 2 weeks(sc q2wk), 66 to ACZ885 300 mg sc q2wk, 69 to ACZ885 150 mg sc q4wk, 71 to placebo. 3 were randomized but not treated. All other 274 (98.9%) were treated and had post-baseline efficacy data.
Pre-assignment Details: Enrollment in core & CACZ885A2201E2 was determined by how many entered first extension study. Study protocols did not mandate that patients continue treatment in the extension phase and furthermore the reason for not continuing from the Core to the Extension phase was not capture. A total of 6.6% completed extensions.
Groups:
- Canakinumab 600 mg IV + 300 mg q2wk: Participants received canakinumab 600 mg intravenous (IV) loading dose on Day 1 and 300 mg subcutaneous injections every 2 weeks (q2wk) for 12 weeks in the Core Phase. In the Extension Phase, participants received 300 mg canakinumab every 4 weeks subcutaneously, until a protocol amendment in January 2009 decreased the dose to 150 mg every 4 weeks. Participants in this treatment group who participated in the Extension Phase are represented in the 'Canakinumab 300 mg q2wk' treatment group in the Extension Phase table below.
Period: Core Study
Arm/Group | Canakinumab 600 mg IV + 300 mg q2wk | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Started | 71 | 64 | 69 | 70
Completed | 62 | 56 | 65 | 63
Not Completed | 9 | 8 | 4 | 7
Not completed — Adverse Event | 5 | 3 | 1 | 1
Not completed — Abnormal Laboratory Values | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 3 | 0 | 4
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 2
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0
Not completed — Administrative Problems | 1 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 2 | 0
Period: Extension Phase
Arm/Group | Canakinumab 600 mg IV + 300 mg q2wk | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Started | 0 (Participants are represented in the Canakinumab 300 mg q2wk treatment group.) | 110 (Includes participants who completed the Core phase in the Canakinumab 600 mg IV + 300 mg q2wk group.) | 59 | 58
Completed | 0 | 8 | 4 | 3
Not Completed | 0 | 102 | 55 | 55
Not completed — Adverse Event | 0 | 9 | 5 | 4
Not completed — Lack of Efficacy | 0 | 16 | 14 | 11
Not completed — Withdrawal by Subject | 0 | 5 | 3 | 4
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0
Not completed — Administrative Problems | 0 | 69 | 32 | 35
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Canakinumab 600 mg IV + 300 mg q2wk | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo | Total
Number analyzed (Participants) | 71 | 64 | 69 | 70 | 274
Age, Customized [Number; unit: participants] — Demographics for the Core Study population. The number of patients in the core phase was 274.
  participants
    ≥18 - <41 years | 5 | 5 | 7 | 7 | 24
    ≥41 - <65 years | 50 | 31 | 43 | 43 | 167
    ≥65 - <75 years | 11 | 18 | 16 | 16 | 61
    ≥75 years | 5 | 10 | 3 | 4 | 22
Age, Customized [Number; unit: participants] — Demographics for the Extension study population. The number of participants in the optional extension phase was less than the overall number of baseline participants who started the study. Total number of patients is 227.
  participants
    ≥18 - <41 years | NA — This group did not exist in the extension studies, only in core. | 7 | 6 | 6 | 19
    ≥41 - <65 years | NA — This group did not exist in the extension studies, only in core. | 66 | 39 | 38 | 143
    ≥65 - <75 years | NA — This group did not exist in the extension studies, only in core. | 25 | 12 | 12 | 49
    ≥75 years | NA — This group did not exist in the extension studies, only in core. | 12 | 2 | 2 | 16
Sex: Female, Male [Count of Participants; unit: Participants] — Demographics for the Core Study population.
  Participants
    Female | 60 | 57 | 56 | 52 | 225
    Male | 11 | 7 | 13 | 18 | 49
Gender [Number; unit: participants] — Demographics for the Extension study population. The number of patients in the optional extension phase was less than the overall number of baseline participants who started the study. Total number of patients is 227.
  participants
    Female | 0 | 94 | 47 | 44 | 185
    Male | 0 | 16 | 12 | 14 | 42

OUTCOME MEASURES:

1. Primary Outcome: Percentage of American College of Rheumatology [ACR] 50 Criteria Responders at Week 12
Description: Participants were defined as ACR50 responders if they had at least a 50% improvement from Baseline in both the tender and the swollen 28-joint count, and in at least 3 of the following 5 measures:
  * Patient's pain assessment (assessed using a 100 mm Visual Analog Scale [VAS]);
  * Patient's global assessment of disease activity (VAS 100 mm);
  * Physician's global assessment of disease activity (VAS 100 mm);
  * Patient self-assessed disability (Health Assessment Questionnaire (HAQ) score);
  * Acute phase reactant (high sensitivity C-reactive Protein [hsCRP]).
  Details on each of these components are provided in Outcome Measures 10-16. Participants were considered as non-responders if they failed the ACR50 criteria. Participants who prematurely discontinued due to insufficient therapeutic effect were also considered non-responders.
Time Frame: Baseline and Week 12
Population: The intent-to-treat (ITT) population consisted of all patients as randomized that received at least one dose of study drug and had at least one post-baseline efficacy assessment. The number of patients in the analysis includes those with ACR50 evaluation. Last observation carried forward was applied for all the component variables.
Measure: Number; unit: percentage of participants
Arm/Group | Canakinumab 600 mg IV + 300 mg q2wk | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 71 | 64 | 68 | 70
percentage of participants | 9.9 [0.31 to 2.65] | 23.4 [0.91 to 6.05] | 26.5 [1.12 to 7.05] | 11.4 [NA to NA]

2. Secondary Outcome: Percentage of American College of Rheumatology [ACR] 50 Criteria Responders at Weeks 2, 4 and 8
Description: Participants were defined as ACR50 responders if they had at least a 50% improvement from Baseline in both the tender and the swollen 28-joint count, and in at least 3 of the following 5 measures:
  * Patient's pain assessment (assessed using a 100 mm Visual Analog Scale [VAS]);
  * Patient's global assessment of disease activity (VAS 100 mm);
  * Physician's global assessment of disease activity (VAS 100 mm);
  * Patient self-assessed disability (Health Assessment Questionnaire (HAQ) score);
  * Acute phase reactant (high sensitivity C-reactive Protein [hsCRP]).
  Participants were considered as non-responders if they failed the ACR50 criteria. Participants who prematurely discontinued due to insufficient therapeutic effect were also considered non-responders.
Time Frame: Baseline and Weeks 2, 4 and 8
Population: The intent-to-treat (ITT) population. The number of patients in the analysis includes those with ACR50 evaluation. Last observation carried forward was applied for all the component variables. "N" indicates the number of patients included at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Canakinumab 600 mg IV + 300 mg q2wk | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 71 | 64 | 69 | 70
percentage of participants
  Responders at Week 2 [N=70, 64, 69, 70] | 2.9 | 1.6 | 5.8 | 4.3
  Responders at Week 4 [N=71, 64, 69, 70] | 1.4 | 7.8 | 7.2 | 4.3
  Responders at Week 8 [N=71, 64, 69, 70] | 4.2 | 17.2 | 17.4 | 7.1

3. Secondary Outcome: Percentage of American College of Rheumatology [ACR] 20 Criteria Responders
Description: Participants were defined as ACR20 responders if they had at least a 20% improvement from Baseline in both the tender and the swollen 28-joint count, and in at least 3 of the following 5 measures:
  * Patient's pain assessment (assessed using a 100 mm Visual Analog Scale [VAS]);
  * Patient's global assessment of disease activity (VAS 100 mm);
  * Physician's global assessment of disease activity (VAS 100 mm);
  * Patient self-assessed disability (Health Assessment Questionnaire (HAQ) score);
  * Acute phase reactant (high sensitivity C-reactive Protein [hsCRP]).
  Participants were considered ACR20 non-responders if they failed the ACR20 criteria. Patients who prematurely discontinued the study due to insufficient therapeutic effect were also considered non responders.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: The intent-to-treat (ITT) population. The number of patients in the analysis includes those with ACR20 evaluation. Last observation carried forward was applied for all the component variables. "N" indicates the number of patients included at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Canakinumab 600 mg IV + 300 mg q2wk | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 71 | 64 | 69 | 70
percentage of participants
  Responders at Week 2 [N=70, 64, 69, 70] | 17.1 [1.06 to 4.74] | 29.7 [1.27 to 5.82] | 23.2 [1.37 to 6.18] | 14.3 [NA to NA]
  Responders at Week 4 [N=71, 64, 68, 70] | 29.6 | 37.5 | 39.7 | 20.0
  Responders at Week 8 [N=71, 64, 68, 70] | 35.2 | 43.8 | 42.6 | 27.1
  Responders at Week 12 [N=71, 64, 68, 70] | 43.7 | 48.4 | 50.0 | 28.6

4. Secondary Outcome: Percentage of American College of Rheumatology [ACR] 70 Criteria Responders
Description: Participants were defined as ACR70 responders if they had at least a 70% improvement from Baseline in both the tender and the swollen 28-joint count, and in at least 3 of the following 5 measures:
  * Patient's pain assessment (assessed using a 100 mm Visual Analog Scale [VAS]);
  * Patient's global assessment of disease activity (VAS 100 mm);
  * Physician's global assessment of disease activity (VAS 100 mm);
  * Patient self-assessed disability (Health Assessment Questionnaire (HAQ) score);
  * Acute phase reactant (high sensitivity C-reactive Protein [hsCRP]).
  Participants were considered ACR70 non-responders if they failed the ACR70 criteria. Patients who prematurely discontinued the study due to insufficient therapeutic effect were also considered non responders.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: The intent-to-treat (ITT) population. The number of patients in the analysis includes those with ACR70 evaluation. Last observation carried forward was applied for all the component variables. "N" indicates the number of patients included at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Canakinumab 600 mg IV + 300 mg q2wk | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 71 | 64 | 69 | 70
percentage of participants
  Responders at Week 2 [N=70, 64, 69, 70] | 0.0 [0.27 to 10.71] | 1.6 [0.14 to 7.61] | 0.0 [0.37 to 12.12] | 0.0 [NA to NA]
  Responders at Week 4 [N=71, 64, 69, 70] | 0.0 | 1.6 | 4.3 | 0.0
  Responders at Week 8 [N=71, 64, 69, 70] | 0.0 | 4.7 | 5.8 | 2.9
  Responders at Week 12 [N=71, 64, 69, 70] | 4.2 | 3.1 | 5.8 | 2.9

5. Secondary Outcome: Number of Distinct Responders According to ACR20, ACR50 and ACR70 Criteria at Week 12
Description: To assess differences between the level of clinical response attained and not just whether the patient did or did not achieve a particular level of response, participants were categorized as follows:
  1. Did not attain an ACR20 response;
  2. Attained a 20% but not a 50% response;
  3. Attained a 50% but not a 70% response;
  4. Attained a 70% or greater response.
  A participant was considered as improved according to the ACR20, ACR50 or ACR70 criteria if they had at least a 20, 50 or 70% improvement from Baseline, respectively, in both the tender and the swollen 28-joint count, and in at least 3 of the following 5 measures:
  * Patient's pain assessment (100 mm visual analog scale [VAS]);
  * Patient's global assessment of disease activity (VAS 100 mm);
  * Physician's global assessment of disease activity (VAS 100 mm);
  * Patient self-assessed disability (Health Assessment Questionnaire [HAQ] score);
  * Acute phase reactant (high sensitivity C-reactive Protein [hsCRP]).
Time Frame: Baseline and Week 12
Population: The intent-to-treat (ITT) population. The number of patients in the analysis includes those with ACR evaluation. Last observation carried forward was applied for all the component variables.
Measure: Number; unit: participants
Arm/Group | Canakinumab 600 mg IV + 300 mg q2wk | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 71 | 64 | 68 | 70
participants
  No response | 40 | 33 | 34 | 50
  ACR20 - not ACR50 response | 24 | 16 | 16 | 12
  ACR50 - not ACR70 response | 4 | 13 | 14 | 6
  ACR70 response | 3 | 2 | 4 | 2

6. Secondary Outcome: Change From Baseline in Swollen 28-joint Count
Description: The following 28 joints were assessed by the physician for swelling: metacarpophalangeal I-V (10), thumb interphalangeal (2), hand proximal interphalangeal II-V (8), wrist (2), elbow (2), shoulders (2), and knees (2).
  Least squares means (LSM) were derived from an Analysis of Covariance (ANCOVA) model adjusting for treatment and center with baseline value as a covariate.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: ITT Population, the number of patients included in the analysis at each time point is indicated by "N". Last observation carried forward was utilized.
Measure: Least Squares Mean (Standard Error); unit: swollen joints
Arm/Group | Canakinumab 600 mg IV + 300 mg q2wk | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 71 | 64 | 69 | 70
swollen joints
  Week 2 [N=70, 64, 69, 70] | -2.4 (0.53) | -2.7 (0.56) | -3.1 (0.54) | -2.3 (0.54)
  Week 4 [N=71, 64, 69, 70] | -3.4 (0.55) | -4.0 (0.58) | -4.6 (0.56) | -3.0 (0.56)
  Week 8 [N=71, 64, 69, 70] | -4.0 (0.58) | -4.4 (0.61) | -4.9 (0.59) | -3.3 (0.59)
  Week 12 [N=71, 64, 69, 70] | -4.6 (0.64) | -5.3 (0.67) | -5.2 (0.65) | -3.4 (0.65)

7. Secondary Outcome: Change From Baseline in Tender 28-joint Count
Description: The following 28 joints were assessed by the physician for tenderness: metacarpophalangeal I-V (10), thumb interphalangeal (2), hand proximal interphalangeal II-V (8), wrist (2), elbow (2), shoulders (2), and knees (2).
  Least squares means (LSM) were derived from an Analysis of Covariance (ANCOVA) model adjusting for treatment and center with baseline value as a covariate.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: tender joints
Arm/Group | Canakinumab 600 mg IV + 300 mg q2wk | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 71 | 64 | 69 | 70
tender joints
  Week 2 [N=70, 64, 69, 70] | -3.0 (0.68) | -2.1 (0.71) | -3.6 (0.68) | -3.2 (0.69)
  Week 4 [N=71, 64, 69, 70] | -4.1 (0.77) | -4.0 (0.80) | -5.0 (0.78) | -4.2 (0.78)
  Week 8 [N=71, 64, 69, 70] | -4.6 (0.79) | -4.7 (0.83) | -5.4 (0.80) | -4.7 (0.80)
  Week 12 [N=71, 64, 69, 70] | -4.3 (0.86) | -4.8 (0.90) | -6.3 (0.87) | -4.5 (0.87)

8. Secondary Outcome: Change From Baseline in Patient's Pain Intensity
Description: The patient's assessment of pain was performed using a 100 mm visual analog scale (VAS) ranging from no pain (0) to unbearable pain (100). The distance in mm from the left edge of the scale was measured. A negative change from Baseline score indicates improvement in pain intensity.
  Least squares means (LSM) were derived from an Analysis of Covariance (ANCOVA) model adjusting for treatment and center with baseline value as a covariate.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: ITT Population, only patients with a value at both Baseline and post-baseline are included in the analysis. The number of patients included at each time point is indicated by
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Canakinumab 600 mg IV + 300 mg q2wk | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 71 | 64 | 68 | 70
scores on a scale
  Week 2 [N=70, 64, 68, 70] | -6.7 (2.20) | -8.0 (2.29) | -8.3 (2.23) | -4.2 (2.22)
  Week 4 [N=71, 64, 68, 70] | -9.1 (2.40) | -9.6 (2.52) | -11.4 (2.45) | -5.6 (2.45)
  Week 8 [N=71, 64, 68, 70] | -12.2 (2.66) | -12.5 (2.80) | -14.0 (2.72) | -7.6 (2.72)
  Week 12 [N=71, 64, 68, 70] | -14.2 (2.72) | -15.1 (2.87) | -17.0 (2.78) | -10.5 (2.78)

9. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity
Description: The patient's global assessment of disease activity was performed using a 100 mm visual analog scale (VAS) ranging from no arthritis activity (0) to maximal arthritis activity (100), after the question "Considering all the ways your arthritis affects you, draw a line on the scale for how well you are doing". The distance in mm from the left edge of the scale was measured. A negative change from Baseline score indicates improvement in assessment of disease activity.
  Least squares means (LSM) were derived from an Analysis of Covariance (ANCOVA) model adjusting for treatment and center with baseline value as a covariate.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Canakinumab 600 mg IV + 300 mg q2wk | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 71 | 64 | 68 | 70
scores on a scale
  Week 2 [N=70, 64, 68, 70] | -6.4 (2.12) | -7.5 (2.21) | -7.9 (2.15) | -5.0 (2.15)
  Week 4 [N= 71, 64, 68, 70] | -9.4 (2.28) | -11.2 (2.39) | -12.8 (2.33) | -6.1 (2.33)
  Week 8 [N= 71, 64, 68, 70] | -13.9 (2.63) | -15.7 (2.76) | -13.8 (2.68) | -6.9 (2.68)
  Week 12 [N= 71, 64, 68, 70] | -14.5 (2.61) | -17.5 (2.74) | -17.6 (2.66) | -10.1 (2.66)

10. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity
Description: The physician's global assessment of disease activity was performed using a 100 mm visual analog scale (VAS) ranging from no arthritis activity (0) to maximal arthritis activity (100). To enhance objectivity, the physician was not aware of the specific patient's global assessment of disease activity when performing their own assessment on that patient. The distance in mm from the left edge of the scale was measured. A negative change from Baseline score indicates improvement in assessment of disease activity.
  Least squares means (LSM) were derived from an Analysis of Covariance (ANCOVA) model adjusting for treatment and center with baseline value as a covariate.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Canakinumab 600 mg IV + 300 mg q2wk | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 71 | 64 | 68 | 70
scores on a scale
  Week 2 [N=70, 64, 68, 69] | -13.3 (2.21) | -14.8 (2.34) | -15.2 (2.25) | -9.3 (2.25)
  Week 4 [N=71, 64, 68, 70] | -17.7 (2.40) | -20.1 (2.55) | -20.3 (2.46) | -12.2 (2.45)
  Week 8 [N=71, 64, 68, 70] | -20.8 (2.68) | -22.6 (2.86) | -23.6 (2.75) | -16.5 (2.74)
  Week 12 [N=71, 64, 68, 70] | -21.6 (2.82) | -24.0 (3.01) | -26.4 (2.90) | -17.6 (2.88)

11. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire (HAQ) Score
Description: The patient health assessment questionnaire (HAQ) was used to assess the physical ability and functional status of participants as well as quality of life. The disability dimension consists of 20 multiple choice items concerning difficulty in performing eight common activities of daily living; dressing and grooming, arising, eating, walking, reaching, personal hygiene, gripping and activities. Participants choose from four response categories, ranging from 'without any difficulty' (Score=0) to 'unable to do' (Score=3). The overall score is the average of each of the 8 category scores and ranges from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. A negative change from Baseline score indicates improvement in disability status.
  Least squares means (LSM) were derived from an Analysis of Covariance (ANCOVA) model adjusting for treatment and center with baseline value as a covariate.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: ITT Population, only patients with a value at both Baseline and post-baseline are included in the analysis. The number of patients included at each time point is indicated by "N". Last observation carried forward was utilized.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Canakinumab 600 mg IV + 300 mg q2wk | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 71 | 64 | 69 | 70
scores on a scale
  Week 2 [N=70, 64, 69, 70] | -0.1 (0.04) | 0.0 (0.05) | -0.1 (0.04) | -0.1 (0.04)
  Week 4 [N=71, 64, 69, 70] | -0.1 (0.05) | -0.1 (0.05) | -0.2 (0.05) | -0.1 (0.05)
  Week 8 [N=71, 64, 69, 70] | -0.2 (0.06) | -0.1 (0.06) | -0.2 (0.06) | -0.1 (0.06)
  Week 12 [N=71, 64, 69, 70] | -0.2 (0.06) | -0.2 (0.06) | -0.2 (0.06) | -0.1 (0.06)

12. Secondary Outcome: Change From Baseline in High-sensitive C-Reactive Protein (hsCRP) Levels
Description: HsCRP is a marker for inflammation and was measured from blood samples to identify the presence of inflammation, to determine its severity, and to monitor response to treatment.
  Least squares means (LSMs) were derived from an Analysis of Covariance (ANCOVA) model adjusting for treatment and center with baseline value as a covariate.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Canakinumab 600 mg IV + 300 mg q2wk | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 71 | 64 | 69 | 70
mg/L
  Week 2 [N=69, 64, 67, 70] | -5.6 (1.72) | -5.8 (1.79) | -4.7 (1.75) | -1.7 (1.74)
  Week 4 [N=71, 64, 69, 70] | -5.2 (1.69) | -7.4 (1.78) | -6.5 (1.72) | -1.7 (1.73)
  Week 8 [N=71, 64, 69, 70] | -4.3 (1.72) | -6.9 (1.82) | -3.5 (1.75) | 0.0 (1.77)
  Week 12 [N=71, 64, 69, 70] | -5.6 (1.89) | -3.4 (1.99) | -8.0 (1.92) | -0.7 (1.94)

13. Secondary Outcome: Change From Baseline in Disease Activity Score (DAS) 28
Description: The Disease Activity Score (DAS) 28 is a combined index to measure the disease activity in patients with rheumatoid arthritis, and includes the following variables:
  * The number of swollen and tender joints assessed using the 28-joint count;
  * C-reactive protein (CRP) in mg/L;
  * Patient's global assessment of disease activity measured on a 100 mm visual analog scale.
  The DAS28 score ranges from zero to ten. DAS28 above 5.1 means high disease activity whereas a DAS28 below 3.2 indicates low disease activity. Remission is achieved by a DAS28 lower than 2.6.
  Least squares means (LSMs) were derived from an Analysis of Covariance (ANCOVA) model adjusting for treatment and center with baseline DAS28 value as a covariate.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Canakinumab 600 mg IV + 300 mg q2wk | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 71 | 64 | 68 | 70
scores on a scale
  Week 2 [N=69, 64, 66, 70] | -0.7 (0.11) | -0.7 (0.11) | -0.8 (0.11) | -0.5 (0.11)
  Week 4 [N=71, 64, 68, 70] | -0.9 (0.13) | -1.0 (0.13) | -1.1 (0.13) | -0.7 (0.13)
  Week 8 [N=71, 64, 68, 70] | -1.1 (0.14) | -1.2 (0.15) | -1.2 (0.14) | -0.8 (0.14)
  Week 12 [N=71, 64, 68, 70] | -1.2 (0.15) | -1.3 (0.16) | -1.5 (0.15) | -0.9 (0.15)

14. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate
Description: Erythrocyte sedimentation rate (ESR) indirectly measures how much inflammation is in the body. A higher ESR is indicative of increased inflammation. A negative change from Baseline score indicates improvement.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Canakinumab 600 mg IV + 300 mg q2wk | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 71 | 64 | 69 | 70
mm/hr
  Week 2 [N=68, 64, 67, 69] | -9.0 (12.85) | -8.2 (15.97) | -9.0 (12.43) | -2.9 (11.62)
  Week 4 [N=71, 64, 69, 70] | -9.2 (15.11) | -9.6 (17.43) | -11.8 (14.71) | -2.6 (12.94)
  Week 8 [N=71, 64, 69, 70] | -11.3 (16.28) | -12.3 (16.02) | -12.8 (13.89) | -4.4 (15.65)
  Week 12 [N=71, 64, 69, 70] | -11.2 (18.20) | -11.1 (18.12) | -15.1 (14.96) | -4.1 (16.73)

15. Secondary Outcome: Change From Baseline in Rheumatoid Factor Concentration
Description: Rheumatoid factor (RF) is an autoantibody (antibody directed against an organism's own tissues) that is an indicator of inflammation and rheumatoid arthritis.
Time Frame: Baseline and Weeks 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: kIU/L
Arm/Group | Canakinumab 600 mg IV + 300 mg q2wk | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 71 | 64 | 69 | 70
kIU/L
  Week 4 [N=70, 62, 68, 67] | -6.7 (71.53) | -10.6 (99.36) | -16.1 (144.18) | -0.9 (85.28)
  Week 8 [N=70, 63, 69, 70] | -2.6 (117.30) | 22.7 (134.66) | -57.1 (442.24) | 6.0 (91.51)
  Week 12 [N=70, 64, 69, 70] | 2.0 (135.70) | 29.7 (144.91) | -50.7 (531.68) | 16.9 (110.03)

16. Secondary Outcome: Change From Baseline in Short Form 36 Health Survey (SF-36)
Description: The SF-36 measures the impact of disease on overall quality of life and consists of eight subscales (physical function, pain, general and mental health, vitality, social function, physical and emotional health) which can be aggregated to derive a physical-component summary score and a mental-component summary score. Scores for each subscale range from 0 to 10, and the composite scores range from 0 to 100, with higher scores indicating better health. A positive change from Baseline score indicates improvement in quality of life.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Canakinumab 600 mg IV + 300 mg q2wk | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 71 | 64 | 69 | 70
scores on a scale
  Physical component: Week 2 [N=61, 61, 59, 64] | 1.73 (5.013) | 0.27 (5.648) | 2.85 (4.999) | 2.03 (6.996)
  Physical component: Week 4 [N=65, 62, 63, 67] | 2.71 (6.582) | 2.30 (6.972) | 3.21 (6.406) | 2.43 (7.134)
  Physical component: Week 8 [N=67, 62, 63, 68] | 2.62 (6.528) | 2.75 (7.331) | 4.29 (8.757) | 1.96 (7.464)
  Physical component: Week 12 [N=68, 62, 63, 68] | 4.03 (6.519) | 3.05 (7.847) | 5.73 (8.612) | 2.69 (7.846)
  Mental component: Week 2 [N=61, 61, 59, 64] | 0.56 (8.831) | 2.64 (8.425) | 1.21 (8.486) | 0.63 (9.234)
  Mental component: Week 4 [N=65, 62, 63, 67] | 2.18 (9.660) | 2.75 (11.364) | 2.23 (8.634) | 1.75 (8.331)
  Mental component: Week 8 [N=67, 62, 63, 68] | 2.29 (10.505) | 2.83 (11.760) | 3.04 (9.307) | 1.18 (9.580)
  Mental component: Week 12 [N=68, 62, 63, 68] | 1.44 (9.988) | 3.34 (11.927) | 4.06 (10.952) | 0.35 (9.294)

17. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy- Fatigue (FACIT-F)
Description: The fatigue subscale of the FACIT is a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function. Participants respond to each item on a 5-point Likert-type scale (0 = not at all; 1 = a little bit; 2 = somewhat; 3 = quite a bit; 4 = very much) based on their experience of fatigue during the past 2 weeks. The scale score is computed by summing the item scores, after reversing those items that are worded in the negative direction. FACIT Fatigue subscale scores range from 0 to 52, where higher scores represent less fatigue.
  Least squares means (LSMs) were derived from an Analysis of Covariance (ANCOVA) model adjusting for treatment and center with baseline FACIT-F value as a covariate.
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Canakinumab 600 mg IV + 300 mg q2wk | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 71 | 64 | 69 | 70
scores on a scale
  Week 2 [N=62, 63, 63, 64] | 2.5 (0.90) | 1.6 (0.87) | 3.7 (0.89) | 2.5 (0.89)
  Week 4 [N=66, 64, 66, 67] | 3.8 (0.99) | 3.3 (0.99) | 4.9 (0.98) | 2.1 (1.00)
  Week 8 [N=67, 64, 66, 67] | 4.2 (1.13) | 4.0 (1.15) | 4.6 (1.13) | 2.1 (1.15)
  Week 12 [N=67, 64, 66, 67] | 4.9 (1.14) | 3.8 (1.15) | 5.7 (1.14) | 1.4 (1.16)

18. Primary Outcome: Percentage of American College of Rheumatology [ACR] 20 Criteria Responders During the Extension Phase
Description: Participants were defined as ACR20 responders if they had at least a 20% improvement from Baseline in both the tender and the swollen 28-joint count, and in at least 3 of the following 5 measures:
  * Patient's pain assessment (assessed using a 100 mm Visual Analog Scale [VAS])
  * Patient's global assessment of disease activity (VAS 100 mm)
  * Physician's global assessment of disease activity (VAS 100 mm)
  * Patient self-assessed disability (Health Assessment Questionnaire (HAQ) score)
  * Acute phase reactant (high sensitivity C-reactive Protein [hsCRP]).
  Participants were considered as non-responders if they failed the ACR20 criteria. Participants who prematurely discontinued due to insufficient therapeutic effect were also considered non-responders.
Time Frame: Baseline and Weeks 24, 36, 48, 60, 72, 88, 100, 112 and 124
Population: The Extension Study intent-to-treat (ITT) population consisted of all patients who entered the extension study and who received at least one dose of study drug in the extension studies. The number of patients in the analysis at each time point (N) includes those with ACR20 evaluation data available.
Measure: Number; unit: percentage of participants
Groups:
- Canakinumab 300 mg q2wk: Participants received canakinumab 300 mg subcutaneous injections every 2 weeks (q2wk) for 12 weeks in the Core Phase. In the Extension Phase, participants received 300 mg canakinumab every 4 weeks subcutaneously, until a protocol amendment in January 2009 decreased the dose to 150 mg subcutaneous injection every 4 weeks. Includes participants who received the 600 mg intravenous loading dose on Day 1 of the Core phase.
Arm/Group | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 110 | 59 | 58
percentage of participants
  Week 24 [N=105, 57, 56] | 52.4 | 64.9 | 66.1
  Week 36 [N=100, 48, 49] | 57.0 | 66.7 | 63.3
  Week 48 [N=95, 43, 47] | 66.3 | 81.4 | 72.3
  Week 60 [N=87, 40, 42] | 60.9 | 75.0 | 73.8
  Week 72 [N=66, 34, 27] | 62.1 | 76.5 | 74.1
  Week 88 [N=43, 25, 23] | 67.4 | 72.0 | 82.6
  Week 100 [N=21, 12, 14] | 81.0 | 75.0 | 91.7
  Week 112 [N=13, 8, 6] | 76.9 | 75.0 | 66.7
  Week 124 [N=2, 1, 1] | 100.0 | 100.0 | 100.0
  End of Study Visit [N=103, 53, 54] | 51.5 | 54.7 | 61.1

19. Primary Outcome: Percentage of American College of Rheumatology [ACR] 50 Criteria Responders During the Extension Phase
Description: Participants were defined as ACR50 responders if they had at least a 50% improvement from Baseline in both the tender and the swollen 28-joint count, and in at least 3 of the following 5 measures:
  * Patient's pain assessment (assessed using a 100 mm Visual Analog Scale [VAS])
  * Patient's global assessment of disease activity (VAS 100 mm)
  * Physician's global assessment of disease activity (VAS 100 mm)
  * Patient self-assessed disability (Health Assessment Questionnaire (HAQ) score)
  * Acute phase reactant (high sensitivity C-reactive Protein [hsCRP]).
  Participants were considered as non-responders if they failed the ACR50 criteria. Participants who prematurely discontinued due to insufficient therapeutic effect were also considered non-responders.
Time Frame: Baseline and Weeks 24, 36, 48, 60, 72, 88, 100, 112 and 124
Population: The Extension Study intent-to-treat (ITT) population consisted of all patients who entered the extension study and who received at least one dose of study drug in the extension studies. The number of patients in the analysis at each time point (N) includes those with ACR50 evaluation data available.
Measure: Number; unit: percentage of participants
Arm/Group | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 110 | 59 | 58
percentage of participants
  Week 24 [N=106, 57, 56] | 18.9 | 29.8 | 37.5
  Week 36 [N=100, 48, 49] | 24.0 | 31.3 | 32.7
  Week 48 [N=95, 43, 47] | 34.7 | 48.8 | 34.0
  Week 60 [N=87, 40, 42] | 34.5 | 42.5 | 42.9
  Week 72 [N=66, 34, 27] | 37.9 | 58.8 | 48.1
  Week 88 [N=43, 25, 23] | 39.5 | 44.0 | 52.2
  Week 100 [N=21, 13, 14] | 47.6 | 30.8 | 57.1
  Week 112 [N=13, 8, 6] | 23.1 | 62.5 | 66.7
  Week 124 [N=2, 1, 1] | 50.0 | 100.0 | 100.0
  End of Study Visit [N=103, 53, 54] | 23.3 | 35.8 | 35.2

20. Primary Outcome: Percentage of American College of Rheumatology [ACR] 70 Criteria Responders During the Extension Phase
Description: Participants were defined as ACR70 responders if they had at least a 70% improvement from Baseline in both the tender and the swollen 28-joint count, and in at least 3 of the following 5 measures:
  * Patient's pain assessment (assessed using a 100 mm Visual Analog Scale [VAS])
  * Patient's global assessment of disease activity (VAS 100 mm)
  * Physician's global assessment of disease activity (VAS 100 mm)
  * Patient self-assessed disability (Health Assessment Questionnaire (HAQ) score)
  * Acute phase reactant (high sensitivity C-reactive Protein [hsCRP]).
  Participants were considered as non-responders if they failed the ACR70 criteria. Participants who prematurely discontinued due to insufficient therapeutic effect were also considered non-responders.
Time Frame: Baseline and Weeks 24, 36, 48, 60, 72, 88, 100, 112 and 124
Population: The Extension Study intent-to-treat (ITT) population consisted of all patients who entered the extension study and who received at least one dose of study drug in the extension studies. The number of patients in the analysis at each time point (N) includes those with ACR70 evaluation data available.
Measure: Number; unit: percentage of participants
Arm/Group | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 110 | 59 | 58
percentage of participants
  Week 24 [N=106, 57, 56] | 5.7 | 10.5 | 14.3
  Week 36 [N=100, 48, 49] | 7.0 | 4.2 | 12.2
  Week 48 [N=96, 43, 47] | 10.4 | 9.3 | 6.4
  Week 60 [N=87, 40, 42] | 16.1 | 17.5 | 19.0
  Week 72 [N=66, 34, 27] | 15.2 | 20.6 | 14.8
  Week 88 [N=44, 25, 23] | 15.9 | 16.0 | 17.4
  Week 100 [N=21, 14, 14] | 14.3 | 21.4 | 28.6
  Week 112 [N=13, 8, 6] | 7.7 | 37.5 | 33.3
  Week 124 [N=2, 1, 1] | 50.0 | 100.0 | 0.0
  End of Study Visit [N=103, 54, 54] | 13.6 | 16.7 | 13.0

21. Primary Outcome: Change From Baseline in Disease Activity Score (DAS) 28 During the Extension Phase
Description: The Disease Activity Score (DAS) 28 is a combined index to measure the disease activity in patients with rheumatoid arthritis, and includes the following variables:
  * The number of swollen and tender joints assessed using the 28-joint count;
  * C-reactive protein (CRP) in mg/L;
  * Patient's global assessment of disease activity measured on a 100 mm visual analog scale.
  The DAS28 score ranges from zero to ten. DAS28 above 5.1 means high disease activity whereas a DAS28 below 3.2 indicates low disease activity. Remission is achieved by a DAS28 lower than 2.6
Time Frame: Baseline and Weeks 24, 72 and 112
Population: The Extension Study intent-to-treat (ITT) population consisted of all patients who entered the extension study and who received at least one dose of study drug in the extension studies. At each timepoint, only patients with a value at both Baseline and that timepoint are included (N).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 110 | 59 | 58
scores on a scale
  Week 24 [N=103, 56, 54] | -1.60 (1.171) | -1.82 (1.333) | -1.93 (1.474)
  Week 72 [N=63, 31, 26] | -2.18 (1.302) | -2.58 (1.232) | -2.21 (1.132)
  Week 112 [N=13, 8, 6] | -2.00 (1.110) | -2.73 (1.252) | -2.59 (1.916)
  End of Study Visit [N=100, 52, 49} | -1.83 (1.434) | -1.79 (1.551) | -1.86 (1.621)

22. Secondary Outcome: Number of Distinct Responders According to ACR20, ACR50 and ACR70 Criteria at the End of the Extension Study
Description: To assess differences between the level of clinical response attained and not just whether the patient did or did not achieve a particular level of response, patients were categorized as follows:
  1. Did not attain an ACR20 response;
  2. Attained a 20% but not a 50% response;
  3. Attained a 50% but not a 70% response;
  4. Attained a 70% or greater response.
  A participant was considered as improved according to the ACR20, ACR50 or ACR70 criteria if they had at least a 20, 50 or 70% improvement from Baseline, respectively, in both the tender and the swollen 28-joint count, and in at least 3 of the following 5 measures:
  * Patient's pain assessment (100 mm visual analog scale [VAS]);
  * Patient's global assessment of disease activity (VAS 100 mm);
  * Physician's global assessment of disease activity (VAS 100 mm);
  * Patient self-assessed disability (Health Assessment Questionnaire [HAQ] score);
  * Acute phase reactant (high sensitivity C-reactive Protein [hsCRP]).
Time Frame: Baseline and End of Study (up to 124 weeks)
Population: Extension Study ITT population.
Measure: Number; unit: participants
Arm/Group | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 103 | 53 | 54
participants
  No response | 50 | 24 | 21
  ACR20 - not ACR50 response | 29 | 10 | 14
  ACR50 - not ACR70 response | 10 | 10 | 12
  ACR70 response | 14 | 9 | 7

23. Secondary Outcome: Change From Baseline in Swollen 28-joint Count During the Extension Study
Description: The following 28 joints were assessed by the physician for swelling: metacarpophalangeal I-V (10), thumb interphalangeal (2), hand proximal interphalangeal II-V (8), wrist (2), elbow (2), shoulders (2), and knees (2).
Time Frame: Baseline and Weeks 24, 36, 48, 60, 72, 88, 100, 112 and 124.
Population: The Extension Study ITT population. At each timepoint, only patients with a value at both Baseline and that timepoint are included (N).
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 110 | 59 | 58
swollen joints
  Week 24 [N=105, 58, 55] | -6.04 (4.892) | -5.70 (5.119) | -6.93 (5.300)
  Week 36 [N=100, 49, 49] | -7.12 (4.828) | -6.79 (4.365) | -7.05 (4.726)
  Week 48 [N=95, 44, 47] | -7.72 (4.171) | -7.52 (3.622) | -7.74 (4.454)
  Week 60 [N=89, 40, 43] | -7.69 (4.670) | -7.38 (3.737) | -8.65 (4.825)
  Week 72 [N=66, 35, 27] | -7.41 (5.311) | -7.94 (4.143) | -7.60 (3.678)
  Week 88 [N=44, 25, 22] | -8.38 (4.369) | -7.24 (3.666) | -7.50 (3.389)
  Week 100 [N=21, 13, 14] | -8.29 (4.285) | -8.15 (2.824) | -7.56 (2.974)
  Week 112 [N=13, 8, 6] | -7.39 (5.308) | -9.50 (2.976) | -5.83 (5.636)
  Week 124 [N=2, 1, 1] | -6.50 (0.707) | -16.00 (NA) — Mean based on 1 participant. Standard deviation can not be calculated. | -4.00 (NA) — Mean based on 1 participant. Standard deviation can not be calculated.
  End of Study Visit [N=103, 55, 53] | -6.36 (5.477) | -5.99 (4.937) | -6.67 (6.350)

24. Secondary Outcome: Change From Baseline in Tender 28-joint Count During the Extension Study
Description: The following 28 joints were assessed by the physician for tenderness: metacarpophalangeal I-V (10), thumb interphalangeal (2), hand proximal interphalangeal II-V (8), wrist (2), elbow (2), shoulders (2), and knees (2).
Time Frame: Baseline and Weeks 24, 36, 48, 60, 72, 88, 100, 112 and 124.
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 105 | 58 | 55
tender joints
  Week 24 [N=105, 58, 55] | -6.93 (7.078) | -8.27 (7.555) | -8.49 (7.298)
  Week 36 [N=100, 49, 49] | -7.92 (6.793) | -9.83 (6.459) | -8.95 (7.154)
  Week 48 [N=95, 44, 47] | -8.64 (7.193) | -10.75 (5.948) | -10.05 (6.321)
  Week 60 [N=89, 40, 43] | -8.52 (6.915) | -11.10 (6.484) | -10.76 (6.185)
  Week 72 [N=66, 35, 27] | -8.71 (7.556) | -11.37 (7.436) | -9.56 (4.722)
  Week 88 [N=44, 25, 22] | -10.34 (5.995) | -10.76 (7.184) | -9.98 (4.964)
  Week 100 [N=21, 13, 14] | -8.53 (5.780) | -12.00 (5.307) | -9.08 (4.989)
  Week 112 [N=13, 8, 6] | -8.47 (6.205) | -13.63 (6.435) | -9.17 (5.981)
  Week 124 [N=2, 1, 1] | -9.00 (4.243) | -23.00 (NA) — Mean based on 1 participant. Standard deviation can not be calculated. | -8.00 (NA) — Mean based on 1 participant. Standard deviation can not be calculated.
  End of Study Visit [N=103, 55, 53] | -7.93 (7.857) | -8.43 (8.331) | -8.83 (7.573)

25. Secondary Outcome: Change From Baseline in Patient's Pain Intensity During the Extension Study
Description: The patient's assessment of pain was performed using a 100 mm visual analog scale (VAS) ranging from no pain (0) to unbearable pain (100). The distance in mm from the left edge of the scale was measured. A negative change from Baseline score indicates improvement in pain intensity.
Time Frame: Baseline and Weeks 24, 36, 48, 60, 72, 88, 100, 112 and 124.
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 106 | 57 | 56
scores on a scale
  Week 24 [N=106, 57, 56] | -22.8 (26.44) | -24.1 (25.69) | -20.8 (25.61)
  Week 36 [N=100, 48, 48] | -21.7 (29.00) | -28.2 (22.05) | -24.0 (24.13)
  Week 48 [N=96, 43, 47] | -25.1 (28.08) | -30.6 (21.94) | -21.1 (23.02)
  Week 60 [N=87, 40, 42] | -26.3 (27.09) | -27.8 (25.63) | -30.0 (23.04)
  Week 72 [N=66, 34, 27] | -29.0 (27.42) | -35.2 (26.06) | -26.2 (27.63)
  Week 88 [N=43, 25, 23] | -28.5 (30.42) | -29.0 (30.23) | -32.3 (24.84)
  Week 100 [N=21, 13, 14] | -30.7 (23.60) | -27.6 (26.14) | -32.0 (26.15)
  Week 112 [N=13, 8, 6] | -33.3 (20.38) | -17.5 (25.39) | -31.7 (38.93)
  Week 124 [N=2, 1, 1] | -55.0 (15.56) | -17.0 (NA) — Mean based on 1 participant. Standard deviation can not be calculated. | -24.0 (NA) — Mean based on 1 participant. Standard deviation can not be calculated.
  End of Study Visit [N=103, 53, 54] | -19.1 (28.14) | -21.9 (27.19) | -20.9 (27.45)

26. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity During the Extension Study
Description: The patient's global assessment of disease activity was performed using a 100 mm visual analog scale (VAS) ranging from no arthritis activity (0) to maximal arthritis activity (100), after the question "Considering all the ways your arthritis affects you, draw a line on the scale for how well you are doing". The distance in mm from the left edge of the scale was measured. A negative change from Baseline score indicates improvement in assessment of disease activity.
Time Frame: Baseline and Weeks 24, 36, 48, 60, 72, 88, 100, 112 and 124.
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 105 | 57 | 56
scores on a scale
  Week 24 [N=105, 57, 56] | -23.2 (26.12) | -21.9 (23.21) | -18.6 (24.42)
  Week 36 [N=100, 48, 48] | -22.5 (28.61) | -23.8 (23.11) | -20.0 (25.52)
  Week 48 [N=96, 43, 47] | -25.8 (27.92) | -27.2 (21.44) | -23.6 (25.23)
  Week 60 [N=87, 40, 42] | -27.7 (29.08) | -24.4 (24.23) | -26.5 (25.63)
  Week 72 [N=66, 33, 27] | -28.6 (24.54) | -32.1 (26.56) | -24.1 (32.14)
  Week 88 [N=43, 25, 23] | -28.4 (27.77) | -30.9 (25.59) | -29.2 (23.95)
  Week 100 [N=21, 13, 14] | -34.1 (20.69) | -27.6 (21.85) | -31.9 (24.45)
  Week 112 [N=13, 8, 6] | -29.9 (23.05) | -28.5 (19.01) | -36.8 (38.84)
  Week 124 [N=2, 1, 1] | -59.5 (20.51) | -20.0 (NA) — Mean based on 1 participant. Standard deviation can not be calculated. | -21.0 (NA) — Mean based on 1 participant. Standard deviation can not be calculated.
  End of Study Visit [N=103, 52, 54] | -20.4 (27.93) | -19.7 (26.29) | -18.6 (27.61)

27. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity During the Extension Study
Description: The physician's global assessment of disease activity was performed using a 100 mm visual analog scale (VAS) ranging from no arthritis activity (0) to maximal arthritis activity (100). To enhance objectivity, the physician was not aware of the specific patient's global assessment of disease activity when performing their own assessment on that patient. The distance in mm from the left edge of the scale was measured. A negative change from Baseline score indicates improvement in assessment of disease activity.
Time Frame: Baseline and Weeks 24, 36, 48, 60, 72, 88, 100, 112 and 124.
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 105 | 57 | 55
scores on a scale
  Week 24 [N=105, 57, 55] | -30.9 (23.58) | -36.1 (25.59) | -36.0 (23.94)
  Week 36 [N=98, 48, 48] | -31.1 (22.69) | -41.6 (18.24) | -37.3 (24.17)
  Week 48 [N=93, 43, 47] | -34.3 (22.60) | -45.6 (18.09) | -38.8 (24.99)
  Week 60 [N=89, 40, 43] | -34.9 (23.57) | -41.9 (22.92) | -42.3 (24.00)
  Week 72 [N=66, 34, 27] | -37.7 (25.64) | -44.6 (22.32) | -43.8 (18.34)
  Week 88 [N=42, 25, 22] | -41.9 (23.81) | -44.8 (19.42) | -45.4 (19.00)
  Week 100 [N=21, 12, 13] | -45.2 (18.56) | -42.2 (12.93) | -47.6 (17.04)
  Week 112 [N=13, 8, 6] | -45.2 (22.11) | -51.4 (13.11) | -29.0 (33.15)
  Week 124 [N=2, 1, 1] | -54.5 (0.71) | -49.0 (NA) — Mean based on 1 participant. Standard deviation can not be calculated. | -39.0 (NA) — Mean based on 1 participant. Standard deviation can not be calculated.
  End of Study Visit [N=102, 53, 53] | -25.6 (27.23) | -29.7 (25.95) | -31.8 (29.28)

28. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire (HAQ) Score During the Extension Study
Description: The patient health assessment questionnaire (HAQ) was used to assess the physical ability and functional status of participants as well as quality of life. The disability dimension consists of 20 multiple choice items concerning difficulty in performing eight common activities of daily living; dressing and grooming, arising, eating, walking, reaching, personal hygiene, gripping and activities. Participants choose from four response categories, ranging from 'without any difficulty' (Score=0) to 'unable to do' (Score=3). The overall score is the average of each of the 8 category scores and ranges from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. A negative change from Baseline score indicates improvement in disability status.
Time Frame: Baseline and Weeks 24, 36, 48, 60, 72, 88, 100, 112 and 124.
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 107 | 58 | 56
scores on a scale
  Week 24 [N=106, 58, 56] | -0.241 (0.5430) | -0.304 (0.4895) | -0.239 (0.5142)
  Week 36 [N=99, 49, 48] | -0.266 (0.5418) | -0.347 (0.5066) | -0.302 (0.5511)
  Week 48 [N=96, 44, 47] | -0.322 (0.5446) | -0.324 (0.4988) | -0.293 (0.5375)
  Week 60 [N=86, 40, 42] | -0.347 (0.5552) | -0.419 (0.5819) | -0.425 (0.6047)
  Week 72 [N=65, 34, 27] | -0.398 (0.6047) | -0.441 (0.5849) | -0.449 (0.6338)
  Week 88 [N=44, 25, 23] | -0.472 (0.5985) | -0.440 (0.5218) | -0.451 (0.5823)
  Week 100 [N=21, 13, 14] | -0.613 (0.5504) | -0.298 (0.4692) | -0.563 (0.7448)
  Week 112 [N=13, 8, 6] | -0.538 (0.5410) | -0.406 (0.6640) | -0.542 (0.7100)
  Week 124 [N=2, 1, 1] | -0.938 (0.6187) | -0.625 (NA) — Mean based on 1 participant. Standard deviation can not be calculated. | -1.250 (NA) — Mean based on 1 participant. Standard deviation can not be calculated.
  End of Study Visit [N=101, 54, 54] | -0.260 (0.6051) | -0.322 (0.5724) | -0.291 (0.6259)

29. Secondary Outcome: Change From Baseline in High-sensitive C-Reactive Protein (hsCRP) Levels During the Extension Study
Description: HsCRP is a marker for inflammation and was measured from blood samples to identify the presence of inflammation, to determine its severity, and to monitor response to treatment.
Time Frame: Baseline and Weeks 24, 36, 48, 60, 72, 88, 100, 112 and 124.
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 106 | 58 | 55
mg/L
  Week 24 [N=106, 58, 55] | -4.82 (17.914) | -6.45 (14.556) | -9.59 (18.388)
  Week 36 [N=97, 49, 50] | -7.76 (16.771) | -4.57 (14.393) | 0.50 (71.610)
  Week 48 [N=95, 44, 47] | -5.61 (22.335) | -4.63 (13.521) | -11.04 (20.261)
  Week 60 [N=88, 40, 43] | -6.93 (21.160) | 0.49 (47.139) | -7.04 (18.638)
  Week 72 [N=63, 33, 26] | -9.02 (18.067) | -5.29 (15.219) | -7.70 (18.221)
  Week 88 [N=44, 24, 22] | -8.45 (19.060) | -7.31 (13.035) | -7.65 (18.098)
  Week 100 [N=21, 14, 12] | -7.29 (12.850) | -2.74 (17.273) | -10.74 (24.539)
  Week 112 [N=13, 9, 6] | -5.75 (10.438) | -1.80 (18.838) | -19.33 (35.567)
  Week 124 [N=2, 1, 1] | 4.95 (13.364) | -22.70 (NA) — Mean based on 1 participant. Standard deviation can not be calculated. | 0.20 (NA) — Mean based on 1 participant. Standard deviation can not be calculated.
  End of Study Visit [N=101, 57, 52] | -7.01 (17.934) | -2.94 (15.735) | -9.74 (20.766)

30. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate During the Extension Study
Description: as for outcome 14
Time Frame: Baseline and Weeks 24, 36, 48, 60, 72 and 88.
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Canakinumab 300 mg q2wk | Canakinumab 150 mg q4wk | Placebo
Number analyzed (Participants) | 105 | 58 | 54
mm/hr
  Week 24 [N=105, 58, 54] | -14.9 (17.31) | -18.3 (14.96) | -16.8 (17.10)
  Week 36 [N=95, 46, 48] | -14.5 (18.99) | -13.6 (19.09) | -11.3 (25.94)
  Week 48 [N=91, 42, 47] | -15.6 (20.13) | -16.6 (13.44) | -17.0 (18.81)
  Week 60 [N=85, 39, 43] | -17.2 (19.07) | -15.8 (19.08) | -16.7 (19.09)
  Week 72 [N=64, 34, 26] | -18.6 (17.83) | -15.3 (16.39) | -14.1 (23.10)
  Week 88 [N=42, 24, 23] | -19.7 (17.46) | -13.5 (16.38) | -13.3 (20.89)
  End of Study Visit [N=98, 55, 55] | -14.9 (18.09) | -14.0 (17.51) | -15.9 (18.10)

ADVERSE EVENTS:
Groups:
- ACZ885 600mg iv + 300mg sc q2wk: ACZ885 600mg iv + 300mg sc q2wk
- ACZ885 300mg sc q2wk: ACZ885 300mg sc q2wk
- ACZ885 150mg sc q4wk: ACZ885 150mg sc q4wk
- Placebo: Placebo
Arm/Group | ACZ885 600mg iv + 300mg sc q2wk | ACZ885 300mg sc q2wk | ACZ885 150mg sc q4wk | Placebo
Serious Adverse Events (participants affected / at risk) | 11/71 | 16/64 | 12/69 | 16/70
Other Adverse Events (participants affected / at risk) | 42/71 | 38/64 | 39/69 | 40/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACZ885 600mg iv + 300mg sc q2wk (N=71) | ACZ885 300mg sc q2wk (N=64) | ACZ885 150mg sc q4wk (N=69) | Placebo (N=70)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 1 | 0
Infected epidermal cyst (Infections and infestations) | 1 | 0 | 0 | 0
Meningitis (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tumour marker increased (Investigations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Hand deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 3
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cervical myelopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 0
Thromboangiitis obliterans (Vascular disorders) | 0 | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ACZ885 600mg iv + 300mg sc q2wk (N=71) | ACZ885 300mg sc q2wk (N=64) | ACZ885 150mg sc q4wk (N=69) | Placebo (N=70)
Diarrhoea (Gastrointestinal disorders) | 5 | 6 | 3 | 5
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 4 | 0
Nausea (Gastrointestinal disorders) | 4 | 5 | 1 | 4
Fatigue (General disorders) | 3 | 3 | 3 | 5
Oedema peripheral (General disorders) | 3 | 4 | 4 | 6
Bronchitis (Infections and infestations) | 6 | 6 | 4 | 3
Gastroenteritis (Infections and infestations) | 6 | 2 | 0 | 4
Influenza (Infections and infestations) | 1 | 2 | 4 | 3
Nasopharyngitis (Infections and infestations) | 14 | 12 | 12 | 10
Sinusitis (Infections and infestations) | 5 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 6 | 8 | 5 | 8
Urinary tract infection (Infections and infestations) | 7 | 5 | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 3 | 5 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 3 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 4 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 | 8 | 6 | 7
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 4
Dizziness (Nervous system disorders) | 2 | 2 | 1 | 4
Headache (Nervous system disorders) | 8 | 4 | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 5 | 5
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 4 | 1
Hypertension (Vascular disorders) | 3 | 6 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.